CLINICAL TRIAL: NCT01669278
Title: Evaluation of Office-Based Sheathed Flexible Nasopharyngoscopy: A Randomized Controlled Trial
Brief Title: Evaluation of Office-Based Sheathed Flexible Nasopharyngoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UA-Endo001
Record Dates: First submitted 2012-08-07; First posted 2012-08-20 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Otorhinolaryngologic Diseases
Keywords: sheath; flexible; endoscopy; otolaryngology; office
MeSH Terms: conditions — Otorhinolaryngologic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional flexible nasopharyngolaryngoscopy (No Intervention): No sheath procedure
- Sheath flexible nasopharyngolaryngoscopy (Active Comparator): Flexible nasopharyngolaryngoscopy using endosheath
  Interventions: Device: Endosheath

INTERVENTIONS:
Device: Endosheath — Flexible sheathed nasopharyngolaryngoscopy
  Arms: Sheath flexible nasopharyngolaryngoscopy

SUMMARY:
The processing of standard flexible nasopharyngoscopes is a time-consuming and costly process. The goal of this study is to determine the efficiency and cost-effectiveness of sheathed flexible endoscope in an office setting.

DETAILED DESCRIPTION:
Methods: Randomized, single-blinded, controlled trial

Setting: Office practice of two academic otolaryngologists at a community hospital.

Primary Outcomes: Patient pain and discomfort, Optical quality

Secondary Outcomes: Physician and nursing staff satisfaction

Cost-analysis

Comparison: No-sheath flexible nasopharyngoscopy versus sheathed flexible nasopharyngoscopy

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting to the Otolaryngology-Head and Neck Surgery service with complaints warranting flexible endoscopy

Exclusion Criteria:

* Known sinonasal masses or nasal polyposis
* Unable to complete VAS surveys
* Significant septal deviation
* Unable to tolerate in-office flexible nasopharyngoscopy
* Patients who refuse consent

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Patient pain and discomfort | 1 hour
  Patient Pain and Discomfort i. Patient's reported level of pain based on International Association for the Study of Pain definitions of pain on a 100-mm Visual Analogue Scale ii. Patient's reported level of discomfort on a 100-mm Visual Analogue Scale

SECONDARY OUTCOMES:
Physician and staff satisfaction | 1 week
  Physician and support staff satisfaction with easy and efficiency of sheathed scopes.
Optical quality | 1 hour
  Image quality of flexible endoscopy with or without endosheath.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Allan Ho, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada